CLINICAL TRIAL: NCT05677009
Title: Sustainable Preservation of Essential Oxygen Resources: A Phase 4 Crossover Study of the Efficacy, Tolerability and SpO2 Non-inferiority of the BUFEO System: SAVE O2
Brief Title: Sustainable Preservation of Essential Oxygen Resources: A Phase 4 Crossover Study of the BUFEO System: SAVE O2
Acronym: SAVEO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxfo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BUFEO-0572201
Record Dates: First submitted 2022-06-13; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Oxygen Deficiency; Oxygen Therapy
Keywords: oxygen
MeSH Terms: conditions — Hypoxia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a prospective, unblinded, single-center study examining the safety, efficacy, and tolerability of BUFEO device compared to standard of care in hospitalized, oxygen-dependent subjects. In this single-visit study, each visit is expected to be approximately 120 minutes. The total study duration to complete 20 subjects (10 males and 10 females) is expected to be 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BUFEO vs Standard Condition (Other): In the BUFEO vs Standard Condition arm, the patient will receive both treatments. The order in which the subject receives the treatment will be randomized.
  Interventions: Device: BUFEO system; Other: Standard of Care

INTERVENTIONS:
Device: BUFEO system — In the BUFEO Condition, the subject will receive oxygen through the BUFEO system.
  Other Names: BUFEO Condition
Other: Standard of Care — Standard Condition is the baseline apparatus utilized by the subject at the time of enrollment in the study. In the hospital setting, the supplemental oxygen delivery may come from compressed oxygen cylinders or liquid oxygen and is often delivered through a port in the facility wall at the bedside.
  Other Names: Standard Condition

SUMMARY:
The current methods of oxygen supply administer medicinal oxygen to the patient at a constant flow. Oxygen is being delivered when the patient needs it (at inhalation) and when the patient does not need it (at exhalation and at rest) if the volume of oxygen needs to be adjusted, the clinician typically increases the rate of flow in an effort to increase the oxygen concentration in the air inhaled by the patient. This traditional way of administering oxygen is clinically effective but it also wastes significant amounts of oxygen that the patient never uses.

The BUFEO system addresses this problem by altering the supply of oxygen to an on-demand delivery model, the patient receives oxygen only when needed (during inhalation) and no oxygen is wasted at rest or during exhalation.

The aim of this study is to evaluate, the efficacy, tolerability, and non-inferiority in SpO2 of the BUFEO device in saving oxygen and reaching a target SpO2 rate, in comparison to the standard of care by measuring the volume of oxygen used and the SpO2 reached when administering medical oxygen with the traditional supply method and through BUFEO system to hospitalized, oxygen-dependent subjects with pulmonary pathology.

DETAILED DESCRIPTION:
The BUFEO system is a class 2a device that saves oxygen by altering the supply of oxygen to an on-demand delivery model through the insertion of a reservoir between the oxygen source and the patient. The reservoir accepts oxygen from the pressurized source where it is converted to ambient pressure. The BUFEO reservoir is approximately 1.75 Liters in volume and, once full, a shut-off valve automatically stops the flow of oxygen from the source and continues to hold the oxygen at ambient pressure. The rate of flow to BUFEO from the oxygen cylinder has no bearing on the volume or concentration of oxygen dispensed to the subject; the only change in the oxygen when entering the reservoir bag from the pressurized source is that it becomes ambient pressure. BUFEO is designed to be connected directly to the pressurized source, typically 50 psi in hospital settings. From the reservoir, oxygen is withdrawn on-demand by the patient's inhalation. After a certain volume is withdrawn from the BUFEO reservoir, the valve is triggered to open and refill from the pressurized source. The rate of flow from the pressurized source to BUFEO affects only the rate at which the reservoir refills upon valve opening; it has no effect on the rate of flow to the mask. Only the volume that the subject inhales on their own is dispensed at the rate of inhalation. Similar to continuous oxygen delivery systems, oxygen from the BUFEO reservoir is available to the patient at the start of the next inspiration. Unlike continuous delivery systems, the flow of oxygen to the patient stops upon the start of expiration. As a result, BUFEO's on-demand model of oxygen delivery greatly reduces waste.

In addition to the conservation of oxygen dispensed, BUFEO also provides efficiency by delivering a high concentration of oxygen (99.9%) directly from the reservoir. In contrast to the standard pressurized delivery of oxygen where one titrates the concentration of oxygen upward by increasing the rate of flow, the BUFEO device requires a downward titration to reduce the concentration of oxygen. The dilution can be done by allowing a set amount of room air to be entrained and blend with the oxygen as it flows from the reservoir to the patient's mask or cannula.

Safety Assessments Vital Signs

Vital signs will be recorded during the study at various points.

Physical Exam

All subjects will undergo a brief, focused physical exam at screening that includes an examination of the heart and lungs.

BUFEO device monitoring

BUFEO device is an attachment to the oxygen delivery system that allows for unobstructed, on-demand access to oxygen contained in the device's reservoir. Each BUFEO device has undergone thorough quality control testing at the point of manufacturing. Each BUFEO device will also undergo testing by study staff prior to the delivery of any study assessments or treatment as indicated by instructions in the BUFEO operation manual. The study staff will also ensure that the device is turned on via examination of the device's power switch indicator prior to the delivery of any study assessments or treatment.

Oxygen Monitoring

Subjects will be continuously monitored by study staff during the course of the study. Subjects' oxygenation levels will also be monitored continuously with the use of a pulse oximeter, the results of which will be recorded in the study's source documents.

Data Collection and Management Data Management

Source documents provide evidence for the existence of the study participant and substantiate the integrity of the data collected. Study data will be recorded on the provided study source documents. Study source documents, including the participant's original signed informed consent, will be kept and securely maintained at the research site. The investigator must retain all study records and source documents for the maximum time period required by local regulations. Only study staff will have access to study source documents.

Source documents will be scanned and sent to the sponsor for quality assurance and data analysis. Any queries will be sent to the study team for reconciliation.

All final data will be entered into a secure Excel file using double data entry. A final review and database lock will be completed after all queries have been resolved.

Confidentiality

All information generated in this study is considered confidential and must not be disclosed to any person or entity not directly involved with the study without prior written consent from the sponsor. Identification of study participants will be via subject initials and assigned study numbers. Study numbers will be assigned to all subjects (including those who screen fail) at the time of screening. Any participant records or data transferred to the sponsor will contain only these identifiers.

ETHICS AND RESPONSIBILITIES

This study will be conducted in compliance with the protocol, Good Clinical Practice (GCP), International Conference on Harmonization (ICH) guidelines, and all applicable local regulations. The protocol will receive Institutional Review Board/Ethics Committee approval prior to the initiation of study activities. The investigator is responsible for submitting the protocol and information regarding Serious Adverse Events to the Ethics Committee. All ethics committee correspondence will be kept with the study records.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed Informed Consent; and
* Able to read, speak, and understand Spanish; and
* Target Population - subjects must meet all of the following criteria:

  1. Between the ages of 18 and 70, inclusive; and
  2. Hospitalized for a medical condition; and
  3. Prescribed supplemental oxygen of a dose ≥2 Liters/minute by a hospital physician at the time of study screening; and
  4. Utilizing a facemask or nasal cannula (as opposed to ventilator) for delivery of supplemental oxygen at the time of study screening; and
  5. Dependent on supplemental oxygen by demonstrating ≥ 3% reduction (absolute value) in blood oxygenation from baseline within 3 minutes of breathing non-oxygen enriched air (i.e. room air); and
* Willingness to follow all study directions including refraining from activities such as making conversation, telephone calls, eating, sleeping, etc. during the study period.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

* Currently pregnant by self-report; or
* ≤ 72 hours post myocardial infarction; or
* Admitted for the treatment of a hemorrhagic or embolic cerebrovertebral accident (stroke); or
* Baseline Dyspnea NRS Rating of ≥ 8; or
* Exhibiting unstable medical conditions at screening as evidenced by:

  1. Blood oxygen saturation outside of target range, defined as <88% or >92% for patients determined to be hypercapnic, or <92% or >96% for patients determined to be NOT hypercapnic; or
  2. Heart rate either < 50 beats per minute or > 100 beats per minute; or
  3. Systolic blood pressure either < 90 mm Hg or > 180 mm Hg; or
  4. Diastolic blood pressure either < 50 mm Hg or > 100 mm Hg; or
  5. Respiratory rate either < 10 or > 28 per minute; or
  6. Temperature > 38.2 C; or
* Difficulty obtaining / recording pulse oximetry measurements from a finger at screening; or
* Any reason(s) determined by the Investigator that may interfere with subject's ability to participate in study activities, may jeopardize the participant's safety or may jeopardize the quality and integrity of the data. This includes:

  1. The participant is unable to give informed consent or follow instructions during their participation in the study.
  2. The participant had any type of surgery in the past 72 hours and the Investigators do not consider the participant to be in stable condition.
  3. The Investigators anticipate failure to adequately titrate the patient to the target blood oxygen saturation for any reason
  4. Any other reason(s) determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
SpO2 Analysis | from date of screening through visit completion or early termination up to 60 minutes
  The ability of the BUFEO device to maintain blood oxygenation levels comparable to standard, continuous oxygen delivery will be assessed through the use of continuous pulse oximetry recorded every 1 minute by the study staff on the paper data forms, as well as every 2 seconds digitally by the oximeter during BUFEO Condition and Standard Condition. The average and standard deviation of these recorded SpO2 values from minute 0 to 20 (20 minutes total) will be documented for data analysis of the primary endpoint. Total time in and out of the target range will be calculated for the 20-minute total duration.
Quantitative Oxygen Consumption Analysis | from date of randomization until visit completion or early termination up to 60 minutes
  The study will use the Digital Gas Mems Mass Flow Meter Model Mf5712 (0-200 L/min; 0.8 MPa; Siargo, Ltd.) to measure and monitor in-line mass flow rate of oxygen for both study conditions. Total volume from minute 0 to minute 20 will be used in data analyses for the BUFEO Condition and Standard Condition, after the 3-minute stabilization period to allow subjects to acclimate to the new mask or cannula and apparatus of each condition.

SECONDARY OUTCOMES:
Patient-reported dyspnea | from date of screening through visit completion or early termination up to 60 minutes
  Tolerability will be assessed with use of the Dyspnea Numeric Rating Scale (NRS). The Dyspnea NRS will be shown to the subject in printed form, and read aloud verbally to elicit a verbal response from the subject, which will be recorded. The Dyspnea NRS asks "How short-of-breath is the participant right now?" This 11-point scale is anchored at 0- "none at all" and 10- "worst shortness of breath imaginable".
Patient-reported discomfort | from date of screening through visit completion or early termination up to 60 minutes
  Discomfort will be assessed with use of the Discomfort Numeric Rating Scale (NRS). The Discomfort NRS will be shown to the subject in printed form, and read aloud verbally to elicit a verbal response from the subject, which will be recorded. The Discomfort NRS asks "How much discomfort does the participant feel right now breathing through this mask?" This 11-point scale is anchored at 0- "no discomfort at all" and 10-"worst discomfort imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bazoberry, MD, Study Director — Director; Susana Osorno, MD, Principal Investigator — Principal Investigator
Locations (1):
- Hospital Alma Máter de Antioquia, Medellín, Antioquia, Colombia